CLINICAL TRIAL: NCT06400758
Title: Impact/Interest of a Collective Prevention Intervention in Sexual and Emotional Health Among High School Students in Lower Normandy
Brief Title: Impact/Interest of a Collective Prevention Intervention in Sexual and Emotional Health
Acronym: Impex
Status: Completed | Type: Observational
Sponsor: Pole Sante Grace de Dieu (Other)
Responsible Party: Sponsor
Other Study IDs: 20240205
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Public Health
Keywords: prevention; sexual health; students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: questionary — A questionnaire, based on the main sexual health topics frequently discussed, was given to students by the school management prior to an intervention.
  The preventive intervention consisted of comprehensive prevention on the emotional and sexual lives of adolescents. It was carried out by health professionals and was based on questions from the students, who were able to leave their questions anonymously in a box in the school infirmary for several months.
  These questions were collected and used to identify several themes for discussion:
  emotional life, with notions of affection, love, friendship and the notion of "normality", as well as consent and sexual violence physical and sexual aspects, with reminders of the menstrual cycle, contraception, sexually transmitted infections, pregnancy and abortion.
  The same questionnaire was given to students after the intervention, to check whether the prevention intervention had improved their general knowledge.

SUMMARY:
Main objective To measure the effects of a group prevention intervention on the sexual and affective knowledge of high school students in the Basse-Normandie region.

Secondary objective Take stock of what is known about the sexual and emotional health of teenagers.

DETAILED DESCRIPTION:
With the average age at first sexual intercourse in France being 17.6 for girls and 17.2 for boys, according to the 2010 health barometer, sexuality education and prevention seem essential at this age, and upstream.

An Australian qualitative study of young men aged 18 to 24 revealed that the main obstacles to discussing sexual health in general practice included the possibility of embarrassment and the fact that the subject was private. Most said they would only talk to their doctor about a sexual problem if it was very important or urgent: if not, they would prefer to wait for the doctor to initiate the subject.

Sexual health prevention initiatives are therefore essential outside the general practitioner's office, and have been shown to be effective in high schools. This is why the PSLA de la Grâce de Dieu has initiated sexual and emotional health prevention initiatives for students at a high school in Caen.

It therefore seemed interesting to assess these students' knowledge of sexual and emotional health before the PSLA's intervention in the amphitheatre with the students, and then after the intervention, in order to find out whether this large-scale prevention action had an impact on these students' knowledge, in the short and medium term.

ELIGIBILITY:
Inclusion Criteria:

* school students in the 2023-2024 school year

Exclusion Criteria:

* A newsletter was sent to the school's head teachers, the students' parents and the students themselves, informing them of the possible use of the data for research purposes, and the possibility of objecting. The principal teachers provided information on the non-obligation to respond during the distribution of the questionnaires. Students who did not respond to the questionnaire were therefore not included.

Ages: 15 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Intervention in a school setting. This intervention is part of a biology course (Life and Earth Sciences). It is a class project. Theoretically, all high school students are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Rate of knowledge improvement between before and after the intervention | 1 year
  the accuracy of correct answers between before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- PSLA GDD, Caen, France

IPD SHARING:
Plan to Share IPD: No